CLINICAL TRIAL: NCT00414908
Title: A Study to Investigate the Effect of Delayed Release Pancrelipase on Maldigestion in Patients With Exocrine Pancreatic Insufficiency Due to Chronic Pancreatitis and Pancreatectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Gregor Eibes, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S245.3.124; 2004-000227-15 (EudraCT Number)
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Results first posted 2009-09-16 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Pancreatitis; Pancreatectomy; Pancreatic Exocrine Insufficiency
Keywords: Chronic Pancreatitis; Pancreatectomy; Pancreatic Exocrine Insufficiency
MeSH Terms: conditions — Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental)
  Interventions: Drug: Pancrelipase delayed release capsule
- B (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Pancrelipase delayed release capsule — 24,000 unit capsule
  Arms: A
Drug: Placebo Comparator — Placebo
  Arms: B

SUMMARY:
This study assessed the effect of pancrelipase delayed release capsules on fat and nitrogen absorption in subjects with PEI due to Chronic Pancreatitis and Pancreatectomy. There was a run-in with a 5-day of single-blind placebo treatment, followed by a 7-day Double-blind period and a 6-month Open-Label Follow-up.

ELIGIBILITY:
Inclusion Criteria:

Pancreatic exocrine insufficiency has to be proven (in medical history) by the following criteria:

* Direct or indirect pancreatic function test (except stool fat excretion) or Clinical signs of severe steatorrhoea that resolved upon administration of pancreatic supplementation.
* Total stool fat > 40 g over 4 days (using Van De Kamer method)
* Proven chronic pancreatitis
* Females of child-bearing potential must agree to continue using a medically acceptable method of birth control

Exclusion Criteria:

* Ileus or acute abdomen
* Any type of malignancy involving the digestive tract in the last 5 years
* Presence of pseudo-pancreatic cyst ≥ 4
* Continued excessive intake of alcohol or drug abuse
* Known infection with HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (30):
- United States (23):
  - Site 9, Scottsdale, Arizona
  - Site 22, Bristol, Connecticut
  - Site 7, Tampa, Florida
  - Site 6, Atlanta, Georgia
  - Site 17, Chicago, Illinois
  - Site 30, Maywood, Illinois
  - Site 14, Indianapolis, Indiana
  - Site 15, Kansas City, Kansas
  - Site 16, Lexington, Kentucky
  - Site 12, New Orleans, Louisiana
  - Site 3, Boston, Massachusetts
  - Site 2, Ann Arbor, Michigan
  - Site 29, Grand Rapids, Michigan
  - Site 1, Tupelo, Mississippi
  - Site 5, St Louis, Missouri
  - Site 8, Cedar Knolls, New Jersey
  - Site 20, Boone, North Carolina
  - Site 4, Rutherford College, North Carolina
  - Site 10, Cincinnati, Ohio
  - Site 11, Cleveland, Ohio
  - Site 21, Pittsburgh, Pennsylvania
  - Site 13, Dallas, Texas
  - Site 18, Richmond, Virginia
- Site 23, Sofia, Bulgaria
- Site 27, Warsaw, Poland
- Site 19, San Juan, Puerto Rico
- Site 25, Saint Petersburg, Russia
- Site 26, Belgrade, Serbia
- Site 24, Cape Town, South Africa
- Site 28, Kiev, Ukraine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in centers in Bulgaria, Poland, Russia, Serbia, Ukraine and US between April 2007 and August 2008. This report presents the double-blind (DB) period of the study as well as the Open Label (OL) results.
Pre-assignment Details: There was a run-in with a 5-day of single-blind placebo treatment. One hundred and eighty subjects were consented and 179 entered the run-in. A total of 54 subjects were randomly allocated to treatment. Only two subjects did not complete the DB period of the treatment because of protocol violation. Fifty one patients entered the OL period.
Groups:
- Pancrelipase (DB): Pancrelipase delayed release capsules given during the Double-Blind period
- Placebo (DB): Placebo group given during the Double-Blind period
Period: Overall Study
Arm/Group | Pancrelipase (DB) | Placebo (DB)
Started | 25 | 29
Completed | 24 | 28
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pancrelipase (DB) | Placebo (DB) | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 27 | 50
  >=65 years | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 51.7 (9.7) | 50.4 (7.8) | 51.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 18 | 19 | 37
Region of Enrollment [Number; unit: participants]
  Serbia | 1 | 3 | 4
  United States | 6 | 6 | 12
  Poland | 7 | 7 | 14
  Ukraine | 3 | 4 | 7
  Russian Federation | 2 | 2 | 4
  Bulgaria | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change of Coefficient of Fat Absorption (CFA) (%) Between Baseline and End of Double-blind (DB) Period.
Description: The CFA is calculated from fat intake and fat excretion : 100*[fat intake-fat excretion]/fat intake. Higher values indicated a better response.
  Change is calculated as (DB CFA-Baseline CFA).
Time Frame: End of double-blind period (5-7 days)
Population: The analysis was done on the Full Analysis sample. Full Analysis Population consists of all subjects who were allocated to the treatment and had data for at least one post-baseline assessment of any efficacy measurement.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Pancrelipase (DB) | Placebo (DB)
Number analyzed (Participants) | 22 | 27
Percentage | 31.93 (18.57) | 8.72 (12.44)
Statistical Analysis 1: Comparison: Pancrelipase (DB) vs Placebo (DB); The following null hypothesis was tested (μ0 and μ1 denote the treatment group means respectively in the placebo and pancrelipase delayed release capsules group): H0: μ0 = μ1 (i.e., placebo and pancrelipase delayed release capsules are equal). The hypothesis corresponded to the primary objective to show superior efficacy of pancrelipase delayed release capsules over placebo. A non-parametric ANCOVA was used because the necessary assumptions were not met for the parametric ANCOVA; Test type: Superiority or Other; p < 0.0001, Non parametric ANCOVA

2. Secondary Outcome: Change of Coefficient of Nitrogen Absorption (CNA) (%) Between Baseline and End of Double-blind (DB) Period.
Description: The CNA is calculated from nitrogen intake and nitrogen excretion : 100*[nitrogen intake-nitrogen excretion]/nitrogen intake. Higher values indicated a better response. Change is calculated as (DB CNA-Baseline CNA).
Time Frame: End of double-blind period (5-7 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Pancrelipase (DB) | Placebo (DB)
Number analyzed (Participants) | 22 | 27
Percentage | 35.23 (29.05) | 8.85 (28.04)
Statistical Analysis 1: Comparison: Pancrelipase (DB) vs Placebo (DB); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, Non parametric ANCOVA

3. Secondary Outcome: Change From Baseline of Stool Fat (g) Between Baseline and End of Double-blind (DB) Period.
Description: Total amount of fat excreted during the stool collection period. Lower values indicate a better response. Change was calculated as (DB Stool fat - Baseline stool fat).
Time Frame: End of double-blind period (5-7 days)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Grammes
Arm/Group | Pancrelipase (DB) | Placebo (DB)
Number analyzed (Participants) | 22 | 27
Grammes | -147.08 (12.71) | -34.62 (11.47)
Statistical Analysis 1: Comparison: Pancrelipase (DB) vs Placebo (DB); The following null hypothesis was tested (μ0 and μ1 denote the treatment group means in the placebo and pancrelipase delayed release capsules group): H0: μ0 = μ1 (i.e., placebo and pancrelipase capsules are equal). The hypothesis was to show superior efficacy of pancrelipase delayed release capsules over placebo. For this secondary efficacy variable, an analysis of covariance (ANCOVA) model was assumed with the treatment group as a fixed factor and the Stool fat at baseline as a covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Means difference = -112.45, 95% CI [-147.04 to -77.87]

4. Secondary Outcome: Change From Baseline of Stool Nitrogen (g) Between Baseline and End of Double-blind (DB) Period.
Description: Total amount of nitrogen excreted during the stool collection period. Lower values indicate a better response. Change was calculated as (DB Stool nitrogen - Baseline stool nitrogen).
Time Frame: End of double-period (5-7 days)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Grammes
Arm/Group | Pancrelipase (DB) | Placebo (DB)
Number analyzed (Participants) | 22 | 27
Grammes | -17.55 (2.06) | -5.87 (1.85)
Statistical Analysis 1: Comparison: Pancrelipase (DB) vs Placebo (DB); The following null hypothesis was tested (μ0 and μ1 denote the treatment group means in the placebo and pancrelipase delayed release capsules group): H0: μ0 = μ1 (i.e., placebo and pancrelipase capsules are equal). The hypothesis was to show superior efficacy of pancrelipase delayed release capsules over placebo. For this secondary efficacy variable, an analysis of covariance (ANCOVA) model was assumed with the treatment group as a fixed factor and the Stool nitrogen at baseline as a covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Means difference = -11.68, 95% CI [-17.30 to -6.06]

5. Secondary Outcome: Change of Stool Frequency Between Baseline and End of Double-blind (DB) Period
Description: Stool frequency is the average of the daily number of stools recorded during the treatment period. Lower values indicate a better response. Change was calculated as (DB stool frequency - Baseline Stool frequency).
Time Frame: End of double-period (5-7 days)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number
Arm/Group | Pancrelipase (DB) | Placebo (DB)
Number analyzed (Participants) | 23 | 28
Number | -0.55 (0.19) | 0.20 (0.17)
Statistical Analysis 1: Comparison: Pancrelipase (DB) vs Placebo (DB); The following null hypothesis was tested (μ0 and μ1 denote the treatment group means in the placebo and pancrelipase delayed release capsules group): H0: μ0 = μ1 (i.e., placebo and pancrelipase capsules are equal). The hypothesis was to show superior efficacy of pancrelipase capsules over placebo. For this secondary efficacy variable, an analysis of covariance (ANCOVA) model was assumed with the treatment group as a fixed factor and the Stool frequency at baseline as a covariate; Test type: Superiority or Other; p = 0.005, ANCOVA; LS Means difference = -0.76, 95% CI [-1.27 to -0.24]

6. Secondary Outcome: Abdominal Pain at the End of the Double-blind Period.
Description: 4- point ordinal scale on this symptom from 0 (No Abdominal pain) to 3 (Severe abdominal pain).
Time Frame: End of double-period (5-7 days)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pancrelipase (DB) | Placebo (DB)
Number analyzed (Participants) | 23 | 28
Participants
  0 (None) | 12 | 8
  1 (Mild) | 7 | 12
  2 (Moderate) | 4 | 7
  3 (Severe) | 0 | 1

7. Secondary Outcome: Stool Consistency at the End of the Double-blind Period
Description: 4- point ordinal scale on this symptom from 0 (Hard) to 3 (Watery).
Time Frame: End of double-period (5-7 days)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pancrelipase (DB) | Placebo (DB)
Number analyzed (Participants) | 23 | 28
Participants
  0 (Hard) | 0 | 0
  1 (Formed/Normal) | 11 | 5
  2 (Soft) | 12 | 20
  3 (Watery) | 0 | 3

8. Secondary Outcome: Flatulence at the End of Double-blind Period
Description: 4- point ordinal scale on this symptom from 0 (None) to 3 (Severe).
Time Frame: End of double-period (5-7 days)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pancrelipase (DB) | Placebo (DB)
Number analyzed (Participants) | 23 | 28
Participants
  0 (None) | 6 | 0
  1 (Mild) | 13 | 15
  2 (Moderate) | 4 | 12
  3 (Severe) | 0 | 1

9. Other Pre Specified Outcome: Change of Stool Frequency Between "Original" Baseline and End of Open-label Period (OL)
Description: Stool frequency is the average of the daily number of stools recorded during the OL period. Lower values indicate a better response. Change was calculated as (OL stool frequency - Baseline stool frequency).
Time Frame: 27 weeks
Population: This analysis is done on the Open-Label period of 6 months.
Measure: Mean (Standard Deviation); unit: Number
Groups:
- Pancrelipase (OL): Pancrelipase delayed during Open-label. Dosing is directed by the investigator.
Arm/Group | Pancrelipase (OL)
Number analyzed (Participants) | 47
Number | -0.98 (1.26)
Statistical Analysis 1: Comparison: Pancrelipase (OL); Test type: Superiority or Other; p < 0.001, Paired t-test; Mean difference based on all subjects combined using the paired t-test between baseline and visit 8 or early termination

ADVERSE EVENTS:
Groups:
- Pancrelipase (DB): Pancrelipase delayed release capsules meaning the treatment received during the 7-days double-blind period
- Placebo (DB): Placebo group meaning the treatment received during the 7-days double-blind period
- Pancrelipase (OL): Pancrelipase delayed capsules received by the patients during the 6-month Open Label. The dosing was directed by the investigator.
Arm/Group | Pancrelipase (DB) | Placebo (DB) | Pancrelipase (OL)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/28 | 7/51
Other Adverse Events (participants affected / at risk) | 1/24 | 2/28 | 4/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pancrelipase (DB) (N=24) | Placebo (DB) (N=28) | Pancrelipase (OL) (N=51)
Acute and Chronic Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Lower Limb Fractures and dislocations (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal Burns (Injury, poisoning and procedural complications) | 0 | 0 | 1
Diabetes Mellitus (Incl Subtypes) (Metabolism and nutrition disorders) | 0 | 0 | 2
Diabetic Complication Dermal (Metabolism and nutrition disorders) | 0 | 0 | 1
Parenchymal Lung Disorders NEC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pancrelipase (DB) (N=24) | Placebo (DB) (N=28) | Pancrelipase (OL) (N=51)
Hyperglycaemic conditions NEC (Metabolism and nutrition disorders) | 1 | 2 | 0
Upper respiratory Tract infections (Infections and infestations) | 0 | 0 | 4

LIMITATIONS AND CAVEATS:
Only treatment emergent events have been presented. They are defined as events started at or after the 1st administration of study medication and includes events started prior to the 1st administration but which worsened after the 1st intake.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At 60 days prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the Site shall provide to Sponsor a copy and allow Sponsor 60 days to review and comment.